CLINICAL TRIAL: NCT01703429
Title: Complementary and Alternative Medicine (CAM) in Multiple Sclerosis. A Prospective Observational Study of a CAM-using Cohort
Brief Title: Complementary and Alternative Care in Multiple Sclerosis
Acronym: CAM Care in MS
Status: Recruiting | Type: Observational
Sponsor: Bastyr University (Other)
Responsible Party: Principal Investigator, Laurie Mischley, Clinical Research Assistant Professor, Bastyr University
Other Study IDs: BU-11A-1296
Record Dates: First submitted 2012-10-03; First posted 2012-10-10 (Estimated); Last update posted 2020-02-11 (Actual); Status verified 2020-02

CONDITIONS: Multiple Sclerosis
Keywords: Multiple Sclerosis; MS; Complementary and Alternative; CAM
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Individuals with MS

SUMMARY:
This is a prospective, observational study designed to describe disease progression, symptom change, quality of life, diet and lifestyle habits, and frequency of adverse events among patients with multiple sclerosis (MS) who use complementary and alternative medicine (CAM). In addition to describing the patterns of CAM use, this study will also identify and describe the positive deviants, those individuals with the highest quality of life and least amount of disease activity. Positive deviants will be compared to controls in order to describe medication, diet, and lifestyle patterns associated with a lack of MS disease progression and high quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of multiple sclerosis (including relapsing remitting MS, secondary progressive MS, primary progressive MS, clinically isolated syndromes (CIS), radiologically-isolated syndromes (RIS), possible MS, or probable MS.
* Age 18-100

Exclusion Criteria:

* Inability to read/write in English
* Inability or unwillingness to complete surveys every six (6) months. (~ 90 min)

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Any individual with multiple sclerosis is invited to participate.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2012-06; Primary Completion 2030-06 (Estimated); Study Completion 2030-06 (Estimated)

PRIMARY OUTCOMES:
"CAM Therapies" survey | 5 years
  This survey has been developed to identify the complementary and alternative therapies most commonly used by individuals with MS. Results will be reported with descriptive statistics.

SECONDARY OUTCOMES:
Modified Expanded Disability Severity Score (EDSS) | 5 years
  The EDSS will be used to capture disease severity and rates of progression in this cohort.

OTHER OUTCOMES:
PROMIS: Global Health | 5 years
  This outcome measure will be used to assess general health and well-being in this CAM using cohort.

CONTACTS AND LOCATIONS:
Overall Officials: Laurie K Mischley, ND, PhD, MPH, Principal Investigator — Bastyr University
Locations (1):
- Bastyr University Clinical Research Center, Kenmore, Washington, United States